CLINICAL TRIAL: NCT07223658
Title: Phase 1/2a, Double-blind, Placebo-controlled, Single and Multiple Dose-escalating Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamic Effects of ARO-DIMERPA in Adult Subjects With Mixed Hyperlipidemia
Brief Title: Study of ARO-DIMERPA in Adult Participants With Mixed Hyperlipidemia
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Arrowhead Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARODIMERPA-1001
Record Dates: First submitted 2025-10-30; First posted 2025-11-03 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Hyperlipidemia; Mixed
MeSH Terms: conditions — Hyperlipoproteinemia Type II

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ARO-DIMERPA (Experimental): ARO-DIMERPA in single or multiple ascending doses
  Interventions: Drug: ARO-DIMERPA
- Placebo (Placebo Comparator): Placebo (normal saline, 0.9%) in single or multiple matching doses
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ARO-DIMERPA — Subcutaneous (SC) injection
  Arms: ARO-DIMERPA
Drug: Placebo — Calculated volume to match active treatment by SC injection
  Arms: Placebo

SUMMARY:
Study to evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD), and effects on low-density lipoprotein cholesterol (LDL-C) and triglycerides (TGs) of single-dose ARO-DIMERPA and multiple doses of ARO-DIMERPA in adult participants with mixed hyperlipidemia.

ELIGIBILITY:
Inclusion Criteria:

* Willing to follow diet counseling as per Investigator judgment based on local standard of care
* Specific fasting TG, LDL-C, and non-high density lipoprotein cholesterol levels at Screening
* Participants of childbearing potential must agree to use highly effective contraception in addition to a condom during the study and for at least 90 days following the end of the study or last dose of study drug, whichever is later; participants must not donate sperm or eggs during the study and for at least 90 days following the end of the study or last dose of study drug whichever is later

Exclusion Criteria:

* Current use or use within last 365 days or within 5-half-lives before Day 1 based on plasma PK, whichever is longer, of any hepatocyte-targeted siRNA
* Current use or use within last 90 days or within 5-half-lives before Day 1 based on plasma PK, whichever is longer, of any antisense oligonucleotide therapy
* Current use or use within last 60 days from Day 1 of any PCSK9 inhibitor monoclonal antibodies (eg, evolocumab or alirocumab)
* Uncontrolled hypertension
* History of bleeding diathesis or coagulopathy
* Current diagnosis of nephrotic syndrome

Note: Additional inclusion/exclusion criteria may apply per protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2025-12-22 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Emergent Adverse Events (TEAEs) | Up to Week 36

SECONDARY OUTCOMES:
Percent Change from Baseline in Fasting LDL-C | Baseline to Week 36
Percent Change from Baseline in Fasting TGs | Baseline to Week 36
Percent Change from Baseline in Serum apoC-III | Baseline to Week 36
Percent Change from Baseline in Serum PCSK9 | Baseline to Week 36
PK of ARO-DIMERPA: Maximum Observed Plasma Concentration (Cmax) | Through 24 hours postdose
PK of ARO-DIMERPA: Time to Maximum Plasma Concentration (Tmax) | Through 24 hours postdose
PK of ARO-DIMERPA: Area Under the Plasma Concentration (AUC) Versus Time Curve From Time Zero to 24 Hours (AUC0-24) | Through 24 hours postdose
PK of ARO-DIMERPA: AUC Versus Time Curve From Time Zero to the Last Quantifiable Plasma Concentration (AUC0-t) | Through 24 hours postdose
PK of ARO-DIMERPA: AUC Versus Time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) | Through 24 hours postdose
PK of ARO-DIMERPA: Apparent Terminal Elimination Half-life (t1/2) | Through 24 hours postdose
PK of ARO-DIMERPA: Apparent Systemic Clearance (CL/F) | Through 24 hours postdose
PK of ARO-DIMERPA: Apparent Terminal-phase Volume of Distribution (Vz/F) | Through 24 hours postdose
PK of ARODIMERPA: Recovery of Unchanged Drug (Ae) in Urine From Time Zero to 24 Hours Postdose | Through 24 hours postdose
PK of ARO-DIMERPA: Percentage of Administered Drug Recovered (Fe) in Urine From Time Zero to 24 Hours Postdose | Through 24 hours postdose
PK of ARO-DIMERPA: Renal Clearance (CLR) | Through 24 hours postdose

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site 1, Christchurch, New Zealand

IPD SHARING:
Plan to Share IPD: No